CLINICAL TRIAL: NCT00001930
Title: NMDA-Receptor Blockade in Huntington's Chorea
Brief Title: Treatment of Huntington's Chorea With Amantadine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990098; 99-N-0098
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Chorea; Huntington's Disease
Keywords: Amantadine; Chorea; Glutamate Antagonist
MeSH Terms: conditions — Chorea; Huntington Disease | interventions — Amantadine

INTERVENTIONS:
Drug: Amantadine

SUMMARY:
Huntington's disease is a chronic disorder passed on through genetic autosomal dominant inheritance. The condition usually begins between the ages of 30 and 50 years and it is characterized by involuntary movements in the face and extremities, (chorea), accompanied by changes in behavior and gradual loss of the mental function. The disease typically ends in a state of disorientation, impaired memory, judgement, and intellect (dementia).

The objective of this study is to test the effectiveness of the drug amantadine for the treatment of chorea associated with Huntington's disease. Amantadine is an antiviral drug that has been used to treat a variety of illnesses including Parkinson's disease. Amantadine works by attaching to special sites called NMDA (N-methyl-D-aspartate) receptors and blocking the normal activity of glutamate there. Glutamate is an amino acid released by brain cells and has been associated with the symptoms of Parkinson's disease.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the acute effects of the putative NMDA-receptor antagonist amantadine on chorea of patients with Huntington's disease (HD). Participants in this study will have mild to moderate HD associated with chorea.

ELIGIBILITY:
All patients will carry a diagnosis of Huntington's disease confirmed by DNA testing.

Patients will have mild to moderate disease with associated significant chorea.

Ability to comply with study requirements and to report on their condition by telephone.

Males and females between the ages of 18 and 82.

No patients with the presence or history of any medical condition that can reasonably be expected to subject the patient to unwarranted risk.

No patients with renal impairment (serum creatinine exceeding the upper limit of normal).

No patients with a history of intolerance to previous exposure to amantadine.

No patients with an MMSE of less than 18/30.

No patients receiving other anti-chorea therapies (such as Haldol). Those receiving other anti-chorea therapies must stop taking these medications for at least 4 weeks prior to the study to be eligible.

No pregnant women.

Patients must practice effective means of birth control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1999-04; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Coyle JT, Schwarcz R. Lesion of striatal neurones with kainic acid provides a model for Huntington's chorea. Nature. 1976 Sep 16;263(5574):244-6. doi: 10.1038/263244a0. No abstract available. PMID 8731
- [Background] Beal MF, Ferrante RJ, Swartz KJ, Kowall NW. Chronic quinolinic acid lesions in rats closely resemble Huntington's disease. J Neurosci. 1991 Jun;11(6):1649-59. doi: 10.1523/JNEUROSCI.11-06-01649.1991. PMID 1710657